CLINICAL TRIAL: NCT00364689
Title: RICE Trial: Rifaximin In Chronic Hepatic Encephalopathy - A Randomized, Controlled Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficult to recruit participants
Sponsor: University of Miami (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060006; 20060298 (Other: WIRB #)
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Hepatic Encephalopathy
Keywords: Encephalopathy, Hepatic; Portosystemic Encephalopathy; Encephalopathy, Hepatocerebral; Encephalopathy, Portal-Systemic; Encephalopathy, Portosystemic; Hepatic Coma; Hepatic Stupor; Hepatocerebral Encephalopathy; Portal-Systemic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin; Lactulose

ARMS (3):
- lactulose given with a placebo (sugar pill) (Experimental)
  Interventions: Drug: Lactulose; Other: Placebo
- lactulose given with rifaximin (Experimental)
  Interventions: Drug: Rifaximin; Drug: Lactulose
- rifaximin given alone (Active Comparator)
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin
  Arms: lactulose given with rifaximin; rifaximin given alone
Drug: Lactulose
  Arms: lactulose given with a placebo (sugar pill); lactulose given with rifaximin
Other: Placebo
  Arms: lactulose given with a placebo (sugar pill)

SUMMARY:
The purpose of this study is to compare the effectiveness of three different treatments for hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis of any cause
2. History of previous admission for acute HE within 12 months of screening and Conn grade 0-1 HE at time of enrollment
3. An Institutional Review Board (IRB/EC) approved informed consent is signed and dated prior to any study-related activities being initiated.
4. Subject is a male or a non-pregnant and non-lactating female. Women of non-childbearing potential or who are practicing adequate birth control are eligible. The investigator is responsible for determining whether the subject has adequate birth control for study participation.
5. Subject is ≥18 years of age.
6. Subject is capable and willing to comply with all study procedures.
7. If the subject has a history of a portal-systemic shunt, shunt placement or revision must be >6 months from Screening for TIPS or a surgical shunt.

Exclusion Criteria:

1. Subject has a significant medical or psychiatric condition which, in the opinion of the Investigator, precludes participation in the study.
2. Subject has a history of allergy or intolerance to lactulose.
3. Subject has a history of allergy or intolerance to rifampin or rifaximin.
4. Subject has participated in an investigational drug or device study within the 30 days prior to study screening.
5. Subject is pregnant or is lactating.
6. Subject shows evidence of ongoing alcohol or drug dependence, in the opinion of the Investigator.
7. Subject has a visual impairment disorder (e.g., glaucoma, diabetic retinopathy, or macular degeneration) or a neurological disease beyond HE that, in the opinion of the Investigator, could impact their performance on neuropsychological assessments and psychometric tests.
8. Subject has any condition or circumstance that would, in the opinion of the Investigator, prevent completion of the study or interfere with analysis of study results, including history of noncompliance with treatments or visits.
9. Subject's current, required medications are on prohibited concurrent medication listing.
10. Hemoglobin < 8.0 at time of screening
11. Severe hypovolemia or electrolyte abnormalities that would be likely to affect mental function (serum sodium less than 120 mEq/L, serum calcium greater than 11 mg/dL) at time of screening
12. Ongoing gastrointestinal bleeding at time of screening
13. Chronic renal insufficiency with a serum creatinine > 3.0 at time of screening
14. History of tuberculosis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chakradhar Reddy, MD, Principal Investigator — University of Miami
Locations (1):
- Center For Liver Diseases - University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants that were assigned to each Arm/Group is not known due to the data for this study no longer being available as the retention period has passed.
Period: Overall Study
Arm/Group | All Participants
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Data collected is no longer available as the retention period has passed.
Groups:
- Lactulose Given With a Placebo (Sugar Pill): Lactulose
  Placebo
- Lactulose Given With Rifaximin: Rifaximin
  Lactulose
- Rifaximin Given Alone: Rifaximin
- Total: Total of all reporting groups
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospitalizations for Hepatic Encephalopathy (HE)
Time Frame: Month 7
Population: Outcome measure data is not reported as the study was terminated due to difficulty with enrolling participants. Collection of data ceased and data analysis was not performed. Data collected is no longer available as the retention period has passed.
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Changes in Psychometric Testing During Study Period
Time Frame: Month 7
Population: as for outcome 1
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Hospitalization Days for All Causes
Time Frame: Month 7
Population: as for outcome 1
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Death or Survival to Liver Transplantation
Time Frame: Month 7
Population: as for outcome 1
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Rate of Adverse Events With Rifaximin Treatment
Time Frame: Month 7
Population: as for outcome 1
Arm/Group | Lactulose Given With a Placebo (Sugar Pill) | Lactulose Given With Rifaximin | Rifaximin Given Alone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Seven months
Description: Data collected for this study are no longer available because the retention period has passed and the data has been destroyed.
Groups:
- All Study Participants: All study participants enrolled in this study.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Outcome measure data is not reported as the study was terminated due to difficulty with enrolling participants. Collection of data ceased and data analysis was not performed. Data collected is no longer available as the retention period has passed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes